CLINICAL TRIAL: NCT00477282
Title: A Phase 3 Study of Safety and Efficacy of Karenitecin Versus Topotecan Administered for 5 Consecutive Days Every 3 Weeks in Patients With Advanced Epithelial Ovarian Cancer
Brief Title: Karenitecin Versus Topotecan in Patients With Advanced Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioNumerik Pharmaceuticals, Inc. (Industry)
Collaborators: Crown Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KTN32313R
Record Dates: First submitted 2007-05-21; First posted 2007-05-23 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Ovarian Cancer
Keywords: Ovarian; Cancer; Advanced Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — cositecan; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Karenitecin (Experimental)
  Interventions: Drug: Karenitecin
- Topotecan (Active Comparator)
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Karenitecin — Karenitecin 1.0mg/m2/day administered as a single daily IV infusion over 60 minutes for 5 consecutive days every 3 weeks (21 days)
  Other Names: BNP1350
  Arms: Karenitecin
Drug: Topotecan — Topotecan 1.5 mg/m2/day administered as a single daily IV infusion over 30 minutes for 5 consecutive days every 3 weeks (21 days)
  Other Names: Hycamtin
  Arms: Topotecan

SUMMARY:
The objective of this study is to assess the safety and efficacy of karenitecin versus topotecan in patients with platinum/taxane-resistant advanced epithelial ovarian cancer. Additionally, this study will assess the ability of karenitecin to extend the time to disease progression, extend the overall survival time, and reduce the incidence and severity of treatment related hematological toxicities in patients with advanced epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed diagnosis of stage III or IV epithelial ovarian cancer
* Have cancer that is resistant to platinum/taxane-based chemotherapy regimens
* Have measurable, progressive disease
* Have an ECOG PS ≤ 2

Exclusion Criteria:

* Have uncontrolled high blood pressure, uncontrolled diabetes mellitus, or other serious underlying medical condition not compatible with study entry.
* Have a life expectancy < 3 months
* Received prior treatment with a camptothecin (topotecan, CPT-11, or investigational camptothecins).
* Received prior treatment with any platinum agent other than cisplatin or carboplatin.
* Received prior radiation therapy to greater than one-third of the hematopoietic sites (one-third of the pelvis and axial skeleton combined).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2007-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | baseline to measured progressive disease

SECONDARY OUTCOMES:
Overall Survival | baseline to date of death from any cause
Incidence of Anemia | Active treatment period (SAEs and on-going treatment-related AEs at end of treatment will be followed until resolution. All other AEs will be followed for up to 30 days after last treatment administration.
Incidence of Neutropenia | Active treatment period (SAEs and on-going treatment-related AEs at end of treatment will be followed until resolution. All other AEs will be followed for up to 30 days after last treatment administration
Incidence of Thrombocytopenia | Active treatment period (SAEs and on-going treatment-related AEs at end of treatment will be followed until resolution. All other AEs will be followed for up to 30 days after last treatment administration

CONTACTS AND LOCATIONS:
Locations (43):
- Hungary (2):
  - Budapest
  - Győr
- Lithuania (2):
  - Kaunas
  - Klaipėda
- Poland (8):
  - Elblag
  - Krakow
  - Lublin
  - Olsztyn
  - Oploe
  - Poznan
  - Szczecin
  - Tarnów
- Romania (8):
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Iași
  - Oradea
  - Sibiu
  - Suceava County
  - Târgu Mureş
- Russia (23):
  - Ulan-Ude, Rep. of Buryatiya
  - Engel's, Saratov Oblast
  - Isvesk, Udmurtiya Republic
  - Arkhangelsk
  - Birobidzhan
  - Khabarovsk
  - Krasnodar
  - Kursk
  - Magnitogorsk
  - Nizhny Novgorod
  - Novosibirsk
  - Orenburg
  - Petrozavodsk
  - Pyatigorsk
  - Ryazan
  - Saint Petersburg
  - Sochi
  - Stavropol
  - Syktyvkar
  - Tambov
  - Ufa
  - Vladimir
  - Vladivostok

REFERENCES:
- See also: MedlinePlus related topic: Ovarian Cancer — http://www.nlm.nih.gov/medlineplus/ovariancancer.html